CLINICAL TRIAL: NCT07014514
Title: Investigation of Sarcopenia Severity in Patients With Parkinson's Disease
Brief Title: Severity of Sarcopenia in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Büşra Seçkinoğulları Korkusuz, Principal Investigator, Ankara University
Other Study IDs: E-59394181-604.01-112205
Record Dates: First submitted 2025-05-30; First posted 2025-06-11 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: sarcopenia; ultrasonography
MeSH Terms: conditions — Parkinson Disease; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Patients with Parkinson's Disease
- Control Group: Healthy individuals with similar demographic characteristics

SUMMARY:
The aim of the study is to examine the severity of sarcopenia in Parkinson's disease patients. Patients between the ages of 40-75 who have been diagnosed with Parkinson's disease by a neurologist and healthy individuals with similar demographic characteristics will be included in the study as a control group. The staging of Parkinson's patients will be done with the Modified Hoehn and Yahr Scale, and the severity of the disease will be done with the Unified Parkinson's Disease Rating Scale. Within the scope of the study, anterior thigh thicknesses of individuals with Parkinson's disease will be evaluated with ultrasonography. Sarcopenia severity will be determined with the ISarcoPRM algorithm using the ultrasonographic evaluations of the individuals. It is planned to include 80 Parkinson's patients in the study. Parkinson's patients between stages 1-3 according to the Modified Hoehn and Yahr Scale will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Score between 24 and 30 on the Mini Mental State Examination
* Be diagnosed with Parkinson's Disease by a neurologist
* Stage 1-3 on the Modified Hoehn and Yahr Scale

Exclusion Criteria:

* Inability to communicate verbally
* Elderly people with severe visual impairment, neurological disorders in addition to Parkinson's and/or congestive heart failure
* Older adults in whom exercise is not recommended

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Among the patients diagnosed with Parkinson's Disease who come to the neurology clinic for routine examination, patients who meet the appropriate inclusion criteria will be evaluated by the Neurology Specialist and included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-10-25 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic Measurement | Baseline
  For sarcopenia evaluation, anterior thigh muscle thickness will be measured by ultrasonography.
Five Times Sit to Stand Test | Baseline
  This test measures the time it takes for an individual to stand up and sit down 5 times as quickly as possible, starting from a sitting position without using their arms.
Hand Grip Strength | Baseline
  In this test, the individual will sit on a chair with their feet flat on the floor. The Jamar Hand Dynamometer will be used for measurement. They will be asked to squeeze the dynamometer firmly with their shoulders adducted and in neutral rotation, their elbows in 90-degree flexion, their forearms neutral and supported, and their wrists neutral. 3 repetitions will be done and the average will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman Korkusuz, PhD, Study Chair — Atılım University; Ayla Fil Balkan, Assoc Prof, Study Chair — Hacettepe University; Gül Yalçın Çakmaklı, Assoc Prof, Study Chair — Hacettepe University; Büşra Seçkinoğulları Korkusuz, PhD, Principal Investigator — Ankara University
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Studenski SA, Peters KW, Alley DE, Cawthon PM, McLean RR, Harris TB, Ferrucci L, Guralnik JM, Fragala MS, Kenny AM, Kiel DP, Kritchevsky SB, Shardell MD, Dam TT, Vassileva MT. The FNIH sarcopenia project: rationale, study description, conference recommendations, and final estimates. J Gerontol A Biol Sci Med Sci. 2014 May;69(5):547-58. doi: 10.1093/gerona/glu010. PMID 24737557
- [Result] Kara M, Kaymak B, Frontera W, Ata AM, Ricci V, Ekiz T, Chang KV, Han DS, Michail X, Quittan M, Lim JY, Bean JF, Franchignoni F, Ozcakar L. Diagnosing sarcopenia: Functional perspectives and a new algorithm from the ISarcoPRM. J Rehabil Med. 2021 Jun 21;53(6):jrm00209. doi: 10.2340/16501977-2851. PMID 34121127